CLINICAL TRIAL: NCT03002493
Title: An Open-Label Phase I Study to Assess the Effect of Rifampicin on the Pharmacokinetics of Eribulin Mesylate (E7389) in Subjects With Advanced Solid Tumors
Brief Title: To Assess the Effect of Rifampicin on the Pharmacokinetics of Eribulin Mesylate in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-E044-111
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2016-02

CONDITIONS: Tumor
Keywords: Rifampicin; Pharmacokinetics; Eribulin Mesylate; E7389; Advanced Solid Tumors; Tumors
MeSH Terms: conditions — Neoplasms | interventions — eribulin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eribulin mesylate + Rifampicin (Experimental)
  Interventions: Drug: Eribulin mesylate; Drug: Rifampicin

INTERVENTIONS:
Drug: Eribulin mesylate — Treatment phase: During Cycle 1, eribulin mesylate was administered as a 2 to 5 minute (min) intravenous (IV) infusion at 1.4 mg/m2 on Day 1 and Day 15 of 21-day cycle. During subsequent cycles, eribulin mesylate administration as a 2 to 5 min IV infusion at 1.4 mg/m2 on Day 1 and Day 8 of a 21-day cycle.
  Extension phase: Eribulin mesylate was administered continuously as a 2 to 5 min IV infusion at 1.4 mg/m2 on Day 1 and Day 8 of 21-day cycles, as long as the Investigator considered eribulin mesylate therapy to be clinically appropriate.
  Other Names: E7389
Drug: Eribulin mesylate
Drug: Rifampicin — Treatment phase: Rifampicin 600 mg was administered orally once a day, from Day 9 to Day 20 of 28-day cycle of Cycle 1.

SUMMARY:
The primary objective of this study was to assess the effect of cytochrome P450 3A4 enzyme (CYP3A4) induction by rifampicin on the pharmacokinetics (PK) of eribulin mesylate following intravenous (IV) administration in participants with advanced solid tumors. The secondary objectives of this study were to assess the safety of eribulin mesylate when co-administered with rifampicin and assess the safety and activity of eribulin mesylate as a single agent.

DETAILED DESCRIPTION:
The study consisted of 3 phases: Pre-Treatment, Treatment, and Extension. Pre-Treatment Phase had 2 periods: Screening and Baseline. Treatment Phase consisted of intensive PK assessment with eribulin mesylate given IV alone on Day 1 followed by eribulin mesylate given IV on Day 15 with rifampicin given orally from Days 9 to 20. Extension Phase allowed eribulin mesylate treatment to continue for participants without progressive disease or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced solid tumors that have progressed following standard therapy or for which no standard therapy exists (including surgery or radiation therapy)
2. Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy and alopecia Grade 2
3. Age greater than or equal to 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
5. Life expectancy of greater than or equal to 3 months
6. Adequate renal function as evidenced by serum creatinine less than or equal to 2.0 mg/dL (less than or equal to 176 umol/L) or calculated creatinine clearance greater than or equal to 40 mL/minute per the Cockcroft and Gault formula
7. Adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limit of normal (ULN) and alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 times the ULN (in the case of liver metastasis less than or equal to 5 times ULN). In the case ALP greater than 3 times the ULN (in the absence of liver metastasis) or greater than 5 times the ULN (in the presence of liver metastasis), and the participant was also known to have bone metastasis, the liver specific ALP were separated from the total and used to assess the liver function instead of the total ALP
8. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L, hemoglobin greater than or equal to 10.0 g/dL or greater than or equal to 6.2 mmol/L (hemoglobin less than 10.0 g/dL or less than 6.2 mmol/L were acceptable if it were corrected by growth factor or transfusion), and platelets greater than or equal to 100 x 109/L
9. Participants were willing and able to comply with the study protocol for the duration of the study
10. Written informed consent were obtained prior to any study-specific screening procedures with the understanding that the participant may withdraw consent at any time without prejudice
11. Females of childbearing potential with a negative serum beta-Human chorionic gonadotropin or a negative urine pregnancy test at Visit 1 (Screening) and prior to starting study drug(s) (Visit 3). Female participants of childbearing potential who agreed to be abstinent or to use a highly effective method of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, intrauterine device [IUD], or have a vasectomised partner) starting prior to starting study drug, throughout the entire study period and for 30 days after the last dose of study drug. Those women using hormonal contraceptives must also have used an additional approved method of contraception (as described previously). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
12. Male participants who were not abstinent or have not undergone a successful vasectomy, who were partners of women of childbearing potential must have used, or their partners must have used a highly effective method of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, IUD) starting prior to starting study drug(s) and throughout the entire study period and for 30 days after the last dose of study drug. Those with partners using hormonal contraceptives must also have used an additional approved method of contraception (as described previously)

Exclusion Criteria:

1. Hypersensitivity to halichondrin B and/or halichondrin B chemical derivatives or a hypersensitivity to rifampicin
2. Prior participation in an eribulin clinical study, even if not previously assigned to eribulin treatment
3. Preexisting neuropathy greater than Grade 2
4. Any of the following treatments within the specified period before eribulin treatment starts:

   1. chemotherapy, radiation or biological therapy within 2 weeks,
   2. hormonal therapy within 1 week with the exception of prostate cancer patients who are on medical castration with a gonadotropin-releasing hormone analog,
   3. any investigational drug within 4 weeks
5. Any medication, dietary supplements or other compounds or substances known to induce or inhibit cytochrome P450 3A4 (CYP3A4) activity at the time the study starts
6. Presence of impaired intestinal absorption
7. Significant cardiovascular impairment such as history of congestive heart failure greater than Grade II (New York Heart Association [NYHA]), unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia
8. Clinically significant electrocardiograms (ECGs) abnormality, including a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval greater than 500 msec)
9. Known positive human immunodeficiency virus (HIV) status
10. Brain or subdural metastases, unless they had completed local therapy and had discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment with eribulin
11. Presence of meningeal carcinomatosis
12. Any history of or concomitant medical condition that, in the opinion of the Investigator, that would have compromise the participant's ability to safely complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Best overall tumor response | From signing of Informed consent until disease progression, undue toxicity, withdrawal by participant, at the discretion of the investigator or up to approximately 8 Months
Area under the concentration-time curve from zero (pre-dose) extrapolated to infinite time (AUC 0-infinity) for eribulin mesylate +/- rifampicin | Day 1 and Day 15 of Cycle 1 (pre-dose, end of infusion, 15 minute (min), and 30 min, 1, 2, 4, 6, 10, 24, 48, 72, 96, 120 and 144 hours after each eribulin administration)
Maximum observed plasma concentration (Cmax) for eribulin mesylate +/- rifampicin | Day 1 and Day 15 of Cycle 1 (pre-dose, end of infusion, 15 min and 30 min, 1, 2, 4, 6, 10, 24, 48, 72, 96, 120 and 144 hours after each eribulin administration)
Area under the concentration-time curve from zero (pre-dose) to time of last quantifiable concentration (AUC 0-t) for eribulin mesylate | Day 1 and Day 15 of Cycle 1 (pre-dose, end of infusion, 15 min and 30 min, 1, 2, 4, 6, 10, 24, 48, 72, 96, 120 and 144 hours after each eribulin administration)
Time of maximum observed plasma concentration (Tmax) for eribulin mesylate | Day 1 and Day 15 of Cycle 1 (pre-dose, end of infusion, 15 min and 30 min, 1, 2, 4, 6, 10, 24, 48, 72, 96, 120 and 144 hours after each eribulin administration)
Half-life (t1/2) for eribulin mesylate | Day 1 and Day 15 of Cycle 1 (pre-dose, end of infusion, 15 min and 30 min, 1, 2, 4, 6, 10, 24, 48, 72, 96, 120 and 144 hours after each eribulin administration)
Clearance (CL) for eribulin mesylate | Day 1 and Day 15 of Cycle 1 (pre-dose, end of infusion, 15 min and 30 min, 1, 2, 4, 6, 10, 24, 48, 72, 96, 120 and 144 hours after each eribulin administration)
Volume of distribution at steady state (Vss) for eribulin mesylate | Day 1 and Day 15 of Cycle 1 (pre-dose, end of infusion, 15 min and 30 min, 1, 2, 4, 6, 10, 24, 48, 72, 96, 120 and 144 hours after each eribulin administration)

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) as a measure of safety | From date of administration of first dose up to 30 days after the last dose of study treatment, up to approximately 8 months.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - University Medical Center Utrecht, Utrecht